CLINICAL TRIAL: NCT01678872
Title: A Long Term Follow-up Study to Evaluate the Safety of RetinoStat® in Patients With Age-Related Macular Degeneration
Brief Title: A Follow-up Study to Evaluate the Safety of RetinoStat® in Patients With Age-Related Macular Degeneration
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Oxford BioMedica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RS1/002/11
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Long Term Follow up (Other): Long Term follow up of patients who received RetinoStat in a previous study.
  Interventions: Drug: RetinoStat

INTERVENTIONS:
Drug: RetinoStat — Long Term Follow up of patients who received RetinoStat in a previous study

SUMMARY:
The purpose of this study is to examine the long term safety of an experimental gene transfer agent, RetinoStat®, designed to treat neovascular age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

* Must have received a subretinal injection of RetinoStat
* Must have been enrolled in Protocol RS1/001/10

Exclusion Criteria:

* Did not receive RetinoStat® as part of the RS1/001/10 protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2012-08; Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | 14 years
  The number of subjects with treatment emergent adverse events.

SECONDARY OUTCOMES:
The change from baseline in BCVA. | 14 years
  The change from baseline in Best Corrective Visual Acuity.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Campochiaro, MD, Principal Investigator — John Hopkins University Hospital
Locations (3):
- United States (3):
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - John Hopkins University Hospital, Baltimore, Maryland
  - Oregon Health & Science University, Portland, Oregon